CLINICAL TRIAL: NCT02798146
Title: The Early Luteal Progesterone Profile in IVF Patients Triggered With hCG - a Pilot Study
Brief Title: Early Luteal Progesterone Profile After hCG Triggering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCKH/CGRH -01-2016
Record Dates: First submitted 2016-06-05; First posted 2016-06-14 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Infertility
Keywords: in-vitro fertilization; luteal phase
MeSH Terms: conditions — Infertility | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hormonal levels (Other): Blood samples are collected for analysis of LH, E2, hCG and progesterone.
  Interventions: Other: blood collection

INTERVENTIONS:
Other: blood collection — Blood samples are collected on the following days after human chorionic gonadotropin (hCG) injection: Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6

SUMMARY:
This pilot-study will help characterize the serum progesterone profiles in IVF patients and correlate progesterone levels to ovarian follicles obtained after stimulation with exogenous gonadotropins.

DETAILED DESCRIPTION:
The early luteal progesterone profile in IVF differs significantly from the progesterone profile of the natural cycle, in which the peak is reached around the time of implantation. With this non-invasive trial investigators wish to further explore the early luteal phase profiles of progesterone and hCG in order to optimize current luteal phase support policies in IVF and hopefully increase ongoing pregnancy rates.

Stimulation, monitoring, and oocyte pick-up will be performed according to the standard procedure of the clinic. On the day of trigger with 5.000 IU hCG a blood sample will be drawn prior to triggering for subsequent analysis. Moreover, all ovarian follicles on each side equal to or above 11 mm will be registered. Oocyte pick-up and timing of the trigger bolus will be performed according to the standard procedures of the unit.

A total 10 blood samples will be drawn during this trial - please see "blood sampling". Blood samples will be collected on the following days for subsequent analysis of LH, E2, hCG and progesterone.

All embryos will be cryo-preserved for transfer in subsequent frozen/thaw embryo transfer cycles.

Primary endpoint Serum concentrations of progesterone, LH, E2, and hCG during early luteal phase.

Secondary endpoints The correlation between follicles ≥ 11 mm and progesterone in early luteal phase

Data are analyzed using SPSS version 20 software. All tests are two tailed, and P<0.05 is considered statistically significant. Continuous variables are presented as mean +/- SD and are tested by student's t-test. Categorical data are expressed as numbers and compared using the Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* IVF patients who meet the following criteria:
* Freeze all cycle after hCG trigger
* Age 18 - 38
* Body Mass Index (BMI) < 28kg/m2
* Normal ovarian reserve, defined by Anti-Mullerian Hormone (AMH) > 1.25 ng/ml or Antral Follicle Count (AFC) ≥ 6 measured within two months prior to stimulation start
* Receiving Gonadotropin Releasing Hormone Antagonist co-treatment during ovarian stimulation
* Agreement to participate in the study, and to disclose any medical events to the investigator. The subject must be willing and able to comply with the protocol requirements for the duration of the study.
* Have given written informed consent with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Previous poor response (≤ 3 oocytes) after high dose FSH stimulation
* Hyper-response defined as >20 follicles ≥ 14 mm
* Chronical medical conditions like Diabetes, Crohns disease, Thyroid disease, Hepatitis B and Sexually Transmitted Diseases Simultaneous participation in an interventional clinical trial.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
change in serum concentrations of progesterone | in 6 days after human chorionic gonadotropin injection
  Blood samples are collected at ten points of time.
change in serum concentrations of luteinizing hormone | in 6 days after hCG injection
  Blood samples are collected at ten points of time.
change in serum concentrations of estradiol | in 6 days after hCG injection
  Blood samples are collected at ten points of time.
change in serum concentrations of hCG | in 6 days after hCG injection
  Blood samples are collected at ten points of time.

SECONDARY OUTCOMES:
number of follicles larger than 11 millimeters | on the day of hCG injection
  Number of follicles are counted on ultrasound image.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vuong LN, Ho TM, Pham TD, Ho VNA, Andersen CY, Humaidan P. The early luteal hormonal profile in IVF patients triggered with hCG. Hum Reprod. 2020 Jan 1;35(1):157-166. doi: 10.1093/humrep/dez235. PMID 31967304